CLINICAL TRIAL: NCT00108784
Title: The Effect of Decreases in Energy Density on Weight Loss and Weight Maintenance
Brief Title: Factors Affecting Caloric Regulation in Human Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FACTORS (completed); R37DK039177 (NIH)
Record Dates: First submitted 2005-04-18; First posted 2005-04-19 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
Keywords: reduced-energy-density diet; fat-restricted diet; fruit; vegetables; ad libitum intake; weight loss; obesity
MeSH Terms: conditions — Obesity; Weight Loss

INTERVENTIONS:
Behavioral: Reduced-energy-density diet

SUMMARY:
This study will test the hypothesis that reducing the energy density of the diet by incorporating more water-rich foods will result in: 1) greater weight loss and weight maintenance; 2) greater diet satisfaction and satiety; and 3) more healthful dietary patterns than reducing dietary fat alone.

DETAILED DESCRIPTION:
Energy density refers to the amount of calories (energy) in a given weight of food. For the same amount of energy, a larger volume (weight) of food can be consumed if the food or diet is low in energy density than if the food or diet is high in energy density. The two nutrients that have the largest impact on energy density are fat and water. Foods high in fat and low in water content are typically high in energy density, whereas foods low in fat and high in water content, such as fruits and vegetables, are low in energy density. This study will examine whether there are increased benefits for weight loss and weight maintenance when the ad libitum consumption of water-rich foods is added to a reduced-fat diet, thus making it even lower in energy density.

Comparisons: Reduced-energy-dense diet and Reduced-fat diet

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* BMI (body mass index) 30 through 40 kg/m2
* Normal blood pressure
* LDL (low density lipoprotein)-cholesterol < 90th percentile recommendations
* Triglycerides, fasting blood glucose, and all other blood values within normal ranges
* Able to participate in low to moderate physical activity.

Exclusion Criteria:

* Heart disease
* Diabetes - type I or II
* High blood pressure
* Renal or kidney disease
* Gastrointestinal disease
* Blood clotting disorder
* Liver disease or cirrhosis
* Any oral steroids
* Gout (requiring treatment)
* Anemia
* Lung disease
* Cancer within the last 5 years
* Thyroid disease

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2003-03; Study Completion 2004-07

PRIMARY OUTCOMES:
Weight loss
Weight maintenance

SECONDARY OUTCOMES:
Changes in diet: quality and patterns, energy density, and fat content
Changes in lipids
Satisfaction with the two different dietary methods for weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Rolls, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- General Clinical Research Center: Penn State University, State College, Pennsylvania, United States

REFERENCES:
- [Background] Rolls BJ, Drewnowski A, Ledikwe JH. Changing the energy density of the diet as a strategy for weight management. J Am Diet Assoc. 2005 May;105(5 Suppl 1):S98-103. doi: 10.1016/j.jada.2005.02.033. PMID 15867904
- [Background] Rolls BJ, Ello-Martin JA, Tohill BC. What can intervention studies tell us about the relationship between fruit and vegetable consumption and weight management? Nutr Rev. 2004 Jan;62(1):1-17. doi: 10.1111/j.1753-4887.2004.tb00001.x. PMID 14995052
- [Background] Bell EA, Rolls BJ. Energy density of foods affects energy intake across multiple levels of fat content in lean and obese women. Am J Clin Nutr. 2001 Jun;73(6):1010-8. doi: 10.1093/ajcn/73.6.1010. PMID 11382653
- [Background] Rolls BJ, Bell EA. Dietary approaches to the treatment of obesity. Med Clin North Am. 2000 Mar;84(2):401-18, vi. doi: 10.1016/s0025-7125(05)70228-5. PMID 10793649
- [Background] Rolls BJ, Bell EA, Thorwart ML. Water incorporated into a food but not served with a food decreases energy intake in lean women. Am J Clin Nutr. 1999 Oct;70(4):448-55. doi: 10.1093/ajcn/70.4.448. PMID 10500012
- [Result] Ello-Martin JA, Roe LS, Ledikwe JH, Beach AM, Rolls BJ. Dietary energy density in the treatment of obesity: a year-long trial comparing 2 weight-loss diets. Am J Clin Nutr. 2007 Jun;85(6):1465-77. doi: 10.1093/ajcn/85.6.1465. PMID 17556681
- See also: Research lab at Penn State University — http://nutrition.hhdev.psu.edu/foodlab/